CLINICAL TRIAL: NCT00385567
Title: A Phase 2 Randomized, Controlled Trial of PEHRG214 in HIV-Infected Patients
Brief Title: A Trial of PEHRG214 in HIV-Infected Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty recruiting eligible patients in timely fashion
Sponsor: Virionyx Corporation Limited (Industry)
Responsible Party: Simon Wilkinson, Virionyx Corporation Limited
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRG2
Record Dates: First submitted 2006-10-01; First posted 2006-10-09 (Estimated); Last update posted 2010-08-26 (Estimated); Status verified 2010-08

CONDITIONS: HIV Infections
Keywords: AIDS; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: PEHRG214

SUMMARY:
HRG2 is a Phase 2 randomized, controlled, open-label, multi-dose trial to determine the efficacy, safety, immunogenicity, and pharmacokinetic profile of PEHRG214 in HIV-infected patients, treated three times weekly for up to 16 weeks.

All patients are receiving optimized standard of care HAART.

The primary objective of the study is to determine the effect of PEHRG214 in decreasing the viral load (>=1.0 log10), as compared to a Control group. The primary hypothesis is that treatment with PEHRG214 will result in clinically meaningful and sustained viral load suppression.

The total sample size is 70-74 patients from approximately 8-10 participating study centers. The first 16-20 patients are enrolled in the non-randomized "pilot arm" and 54 subsequent patients are randomized (2:1 within center) to Treatment or Control group. The total study duration is 7-12 months.

DETAILED DESCRIPTION:
The study design is a randomized, controlled, open-label multi-dose trial of PEHRG214 administered intravenously three times weekly, with the potential for dose escalation in selected patients. Patients with HIV infection, viral load at least 10 times greater than the site laboratory's lower limit of detection and CD4 count of <220 cells/mm3, will be entered into the trial. All patients must be taking an optimized background regimen (OBR) of antiretroviral agents, as confirmed by the Principal Investigator, in accordance with the U.S. Department of Health and Human Services Guidelines for the Use of Antiretroviral Agents in HIV-1 Infected Adults and Adolescents, May 4, 2006.

A non-randomized "pilot arm" of 16-20 patients will first receive 2.0 mg/kg three times weekly for 12 doses. After a "pilot arm" patient has received at least 12 doses of PEHRG214 at 2.0 mg/kg, dose escalation to 4.0 mg/kg three times weekly will follow a scheme based on adverse event, HAGAR, and viral load assessments for each individual patient, and in certain cases, further review by the DSMB. After the "pilot arm" patients have received 12 doses at 4.0 mg/kg, all subsequent patients will enter the protocol at the 4.0 mg PEHRG214/kg level. The subsequent 54 patients will be randomized, in 2:1 ratio within center, to the Treatment group and Control group, respectively. The treatment group will receive PEHRG214 at a dose of 4.0 mg/kg three times weekly for up to 48 doses (16 weeks). The Control group will not receive the investigational drug, but will undergo observation while receiving standard of care HAART.

After at least 12 doses of PEHRG214 at 4.0 mg/kg, dose escalation to 8.0 mg/kg three times weekly will follow a scheme based on adverse event, HAGAR, and viral load assessments for each individual patient, and in certain cases, further review by the DSMB.

The Control patients will be evaluated every 4 weeks for 16 weeks according to the Schedule of Assessments in Appendix 1F. After 16 weeks, these patients will have the option of being enrolled in an extension protocol where they can receive PEHRG214.

ELIGIBILITY:
Inclusion Criteria:

* Serological documentation of HIV infection at any time prior to study entry.
* CD4 cells count of <220 cells/mm3 within 35 days of study drug administration.
* Viral load at least 10 times greater than the site laboratory's lower limit of detection within 35 days of study drug administration.
* The patient must be taking an optimized background regimen (OBR) of antiretroviral agents, as confirmed by the Principal Investigator, in accordance with the US Department of Health and Human Services Guidelines for the Use of Antiretroviral Agents in HIV-1 Infected Adults and Adolescents, May 4, 2006; (http://www.aidsinfo.nih.gov/guidelines/) or comparable standard of care guidelines.
* OBR has been individually selected for the patient based on prior viral resistance testing and antiretroviral treatment history.
* OBR has been stable for at least 4 weeks prior to Screening and is expected to remain stable for the duration of the trial.
* Karnofsky performance status >=60%.
* Adequate laboratory parameters: absolute neutrophil count >1000 cells/mm3 hemoglobin >9.0 g/dL; platelets >75,000/mm3; creatinine <1.5 x upper limit of normal; SGOT/SGPT <3.0 x upper limit of normal; bilirubin <2.0 mg/dL. Note: Patients who are taking indinavir or atazanavir will be allowed on this trial if their bilirubin is >3.0 mg/dL and if it is deemed by both the Principal Investigator and patient's physician that the elevated bilirubin is solely related to indinavir or atazanavir.
* Women of Child Bearing Potential (WOCBP) must have a negative serum or urine pregnancy test.
* Prophylaxis for Pneumocystis carinii pneumonia using aerosolized pentamidine, trimethoprim/sulfamethoxazole, mepron or dapsone is required for study patients.
* Signed informed consent.

Exclusion Criteria:

* Patient is pregnant or lactating.
* Active opportunistic infection which is progressive, or imminently disabling or life-threatening, in the judgment of the Principal Investigator.
* Cytotoxic chemotherapy, interferon treatment, or radiation therapy within the preceding 3 weeks (patients who have received intralesional chemotherapy will not be excluded, however).
* Any investigational drugs within 30 days or any investigational biologic agents within 6 weeks. Patients taking antiretroviral investigational drugs within Expanded Access Programs (21CFR312.34) are not excluded from participation, provided these drugs are not excluded elsewhere in the protocol.
* Patients who have received an HIV vaccine.
* Known hypersensitivity to animal proteins, including red meats, milk, or milk products, or previous treatment with a caprine antibody and HAGAR (Human anti-goat antibody response) or the presence of HAGAR at screening.
* As this is an experimental regimen, patients will not be permitted to enroll if they had been on an effective antiretroviral regimen, which they tolerated well and which they discontinued for the sake of enrolling in this protocol.
* Active drug abuse.
* Any condition which in the Principal Investigator's opinion may render the patient unable to complete the study or which may pose significant risk to the patient.
* Chronic treatment with immunosuppressant drugs, including corticosteroids, except for the treatment of adrenal insufficiency. Topical steroids are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Decrease in viral load >= 1.0 log10 at 16 weeks
Positive changes in CD4 count, weight, and Karnofsky Performance Score at 16 weeks
Improvement in quality of life as determined monthly, using the MOS-HIV Health Survey

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - L.A. Gay & Lesbian Center, Los Angeles, California
  - University of Miami School of Medicine - AIDS Clinical Research Unit, Miami, Florida
  - Northstar Healthcare, Chicago, Illinois
  - University of Iowa - HIV/ AIDS Clinical Trials, Iowa City, Iowa
  - Beth Israel Medical Center - AIDS Clinical Trials Unit, New York, New York
  - University of Texas Southwestern Medical Center - HIV Research Clinic, Dallas, Texas
- Clinical Research Puerto Rico, Inc, San Juan, Puerto Rico

REFERENCES:
- [Background] Verity EE, Williams LA, Haddad DN, Choy V, O'Loughlin C, Chatfield C, Saksena NK, Cunningham A, Gelder F, McPhee DA. Broad neutralization and complement-mediated lysis of HIV-1 by PEHRG214, a novel caprine anti-HIV-1 polyclonal antibody. AIDS. 2006 Feb 28;20(4):505-15. doi: 10.1097/01.aids.0000210604.78385.95. PMID 16470114
- [Background] Dezube BJ, Proper J, Zhang J, Choy VJ, Weeden W, Morrissey J, Burns EM, Dixon JD, O'Loughlin C, Williams LA, Pickering PJ, Crumpacker CS, Gelder FB. A passive immunotherapy, (PE)HRG214, in patients infected with human immunodeficiency virus: a phase I study. J Infect Dis. 2003 Feb 1;187(3):500-3. doi: 10.1086/367710. Epub 2003 Jan 8. PMID 12552435
- [Background] Pett SL, Williams LA, Day RO, Lloyd AR, Carr AD, Clezy KR, Emery S, Kaplan E, McPhee DA, McLachlan AJ, Gelder FB, Lewin SR, Liauw W, Williams KM. A phase I study of the pharmacokinetics and safety of passive immunotherapy with caprine anti-HIV antibodies, (PE)HRG214, in HIV-1-infected individuals. HIV Clin Trials. 2004 Mar-Apr;5(2):91-8. doi: 10.1310/1FLN-8KFC-5HEQ-K19J. PMID 15116285